CLINICAL TRIAL: NCT04965324
Title: Depth of Anaesthesia and Long-term Survival in Elderly Surgical Patients: The Balanced Anaesthesia Study Long-term Follow-up Study
Brief Title: Depth of Anaesthesia and Long-term Survival: The Balanced Anaesthesia Follow-up Study
Acronym: BALANCEDLT
Status: Completed | Type: Observational
Sponsor: Auckland City Hospital (Other Government)
Collaborators: Health Research Council, New Zealand (Other); Australian and New Zealand College of Anaesthetists (Other)
Responsible Party: Sponsor
Other Study IDs: A+9283; ACTRN12612000632897 (Registry Identifier: Australia New Zealand Clinical Trials Registry)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Post-Operative Confusion; Long Term Adverse Effects; Surgery--Complications; Cognitive Dysfunction, Postoperative
Keywords: Anesthesia; Delirium; Incidence; Long Term Survival
MeSH Terms: conditions — Long Term Adverse Effects; Postoperative Cognitive Complications; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anaesthesia Depth BIS 35: BIS 35
  Interventions: Other: Anaesthesia Depth
- Anaesthesia Depth BIS 50: BIS 50
  Interventions: Other: Anaesthesia Depth

INTERVENTIONS:
Other: Anaesthesia Depth

SUMMARY:
Anaesthetic depth and complications after major surgery: an international, randomised controlled trial - The BALANCED trial.

In this large, international, randomised controlled trial that enrolled patients aged 60 years and over with significant comorbidity and at increased risk of complications after major surgery, we found no evidence that light general anaesthesia (bispectral index 50) was superior to deep general anaesthesia (bispectral index 35) in reducing 1-year mortality. The BALANCED long term follow up study will look at whether depth of anesthesia affects long term (beyond 1 year) survival.

The primary hypothesis is that targetting BIS 50 will result in superior long term survival compared to targetting BIS 35.

The two secondary hypotheses are that BIS titration to BIS 50 will

1. reduce local cancer recurrence or metastatic spread and consequently improve long-term survival
2. reduce postoperative delirium and associated cognitive impairment and consequently improve long-term survival

Both these mechanisms would be expected to take longer to manifest as reduced survival than 1-year all-cause mortality primary outcome in the Balanced trial. Trials of cancer outcomes often use 5-year survival or similar timeframes to determine evidence of clinical benefit. A steeper cognitive trajectory due to intermediate outcomes such as delirium and cognitive impairment may take longer than 1 year to produce a clinically important difference in survival 30. The 10.6% relative risk reduction seen in the Balanced trial could translate to a statistically and clinically meaningful survival difference in this high-risk population. This population may have 5-year survival of ~80% translating to an absolute survival difference of ~2% potentially (if the ~10% RRR is maintained beyond 1 year). The alternative is that there is no long-term mortality difference which would provide continuing clinical guidance of the safety of current practice in patients who are not at high risk of delirium. This study could provide a rationale for trials in larger populations (such as the total Balanced trial population) or targeted subgroups such as cancer and delirium to provide further mechanistic insights.

Long-term survival is an important patient-centred outcome. The mechanisms described above may manifest in longer-term outcomes providing a clear rationale for the current trial.

ELIGIBILITY:
Inclusion and exclusion criteria will be the same as the Balanced trial with participants limited to those sites described above. Survival data will be censored at date of accessing mortality database.

Inclusion

1. Age over 60 years and over
2. ASA physical status 3 or 4
3. Surgery expected to last over 2 hours
4. Hospital length of stay expected to be 2 nights or more
5. General anaesthesia with or without major regional block
6. Able to monitor BIS throughout anaesthesia

Exclusion

1. Unable to monitor BIS
2. Unable to consent
3. Surgery with 'wake up' test
4. Propofol infusion for part or all of maintenance of anaesthesia
5. Previous enrolment in Balanced study

Exclusion The intention-to-treat (ITT) population is defined as all randomised participants who met the inclusion and exclusion criteria who had surgery.

The per-protocol (PP) population is defined as all randomised participants in the study who meet all the inclusion/exclusion criteria for BALANCED with BIS group classified according to the actual median BIS value achieved irrespective of randomisation.

Participants were allocated to the BIS=50 group if the achieved median BIS is between 45 and 55 inclusive, and to the BIS=35 group if the achieved median BIS is between 30 and 40 inclusive. Participants who are not within these ranges will be excluded from these analyses.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants who were recruited to the BALANCED Trial and who met the inclusion and no exclusion criteria for analysis of the long term outcome.
Sampling Method: Probability Sample
Enrollment: 6644 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Survival | Between one year and eight years after randomization to the BALANCED Trial
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dr Short, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hopsital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data sharing requests will be assessed by the Balanced Study Steering.Committee.
  Individual, deidentified participant data used in these analyses will be shared 2 years after publication by request from any qualified investigator after approval of a protocol, statistical analysis plan, and receipt of a signed data access agreement via the Research Office of Auckland District Health Board, New Zealand; and after obtaining the approval of the New Zealand Health and Disability Ethics Committees for the project and data release
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 2 years
Access Criteria: Will be available on the clintrials.govt website